CLINICAL TRIAL: NCT00852085
Title: Reducing Youthful Dangerous Driving
Acronym: RYDD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Ted Nirenberg PhD, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R49CE000544-03 (NIH)
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Injuries
Keywords: Counseling; Crime; Adolescent
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group MI (Experimental): Four group counseling sessions and a directed observational visit to the emergency department of a busy urban hospital
  Interventions: Behavioral: Group MI
- Enhanced community service (Active Comparator)
  Interventions: Behavioral: Enhanced community service

INTERVENTIONS:
Behavioral: Enhanced community service — Two educational sessions and volunteering at a local community service site
  Arms: Enhanced community service
Behavioral: Group MI — Four group counseling sessions and two directed observational visits to an emergency department
  Arms: Group MI

SUMMARY:
To examine the effectiveness of four motivational counseling groups and a directed observational experience in the emergency room in comparison to education and community volunteering only, in reducing high risk driving behaviors

ELIGIBILITY:
Inclusion Criteria:

* Age 16-20 years
* Court referred for driving offense
* Speak English

Exclusion Criteria:

* Age over 20 years
* Not court referred
* Not English speaking

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 482 (Actual)
Dates: Start 2005-10; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Rates of traffic offenses | 12 months post intervention completion

SECONDARY OUTCOMES:
Self-reported high risk driving behaviors | 12 months post intervention completion